CLINICAL TRIAL: NCT06686654
Title: A Phase 1/2, Randomized, Observer-blind, Placebo-controlled Multi-arm Study to Evaluate the Safety and Immunogenicity of an hMPV/RSV mRNA Vaccine Candidate in Adult Participants Aged 60 Years and Older
Brief Title: Study of a Human Metapneumovirus/Respiratory Syncytial Virus mRNA Vaccine Candidate Encapsulated in a Lipid Nanoparticle-based Formulation in Adults Aged 60 Years and Older
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VBD00009; U1111-1310-4940 (Other: WHO ICTRP)
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Human Metapneumovirus Immunization; Respiratory Syncytial Virus Immunization
Keywords: hMPV; RSV; respiratory syncytial virus infection; human metapneumovirus infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: Dose-ranging, parallel, multi-center, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stage 1 Sentinel and Main Cohorts: observer-blind; for safety evaluation purposes, the Sponsor Safety Management Team (SMT) will be unblinded for the Sentinel Cohort (including early safety data review [ESDR]) and will be blinded for the Main Cohort.
  Stage 2 Expansion Cohort: observer-blind until all participants complete the Month 6 visit, then open-label Stage 2 Booster Cohort: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- Group A Stage 1 Sentinel Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation A
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group B Stage 1 Sentinel Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation B
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group C Stage 1 Sentinel Cohort (Placebo Comparator): 1 IM injection of placebo
  Interventions: Biological: Placebo
- Group 1 Stage 1 Main Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation C
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 2 Stage 1 Main Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation D
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 3 Stage 1 Main Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation E
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 4 Stage 1 Main Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation F
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 5 Stage 1 Main Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation G
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 6 Stage 1 Main Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation A
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 7 Stage 1 Main Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation B
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 8 Stage 1 Main Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation H
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 9 Stage 1 Main Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation I
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 10 Stage 1 Main Cohort (Experimental): 1 IM injection of investigational hMPV/RSV vaccine formulation J
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 11 Stage 1 Main Cohort (Placebo Comparator): 1 IM injection of placebo
  Interventions: Biological: Placebo
- Group X Stage 2 Expansion Cohort (Experimental): 1 IM injection of selected investigational hMPV/RSV vaccine formulation from Group 1-9 of Stage 1 Main Cohort
  Interventions: Biological: Investigational hMPV/RSV vaccine
- Group 12 Stage 2 Expansion Cohort (Experimental): 1 IM injection of investigational RSV monovalent vaccine
  Interventions: Biological: Investigational RSV vaccine (monovalent)
- Group 13 Stage 2 Expansion Cohort (Experimental): 1 IM injection of investigational hMPV monovalent vaccine
  Interventions: Biological: Investigational hMPV vaccine (monovalent)
- Group 14 Stage 2 Expansion Cohort (Experimental): 1 IM injection of licensed RSV vaccine
  Interventions: Biological: Licensed RSV Vaccine
- Group 15 Stage 2 Booster Cohort (Experimental): 1 IM injection of investigational RSV + hMPV vaccine formulation administered to participants from Group 14 of Expansion Cohort
  Interventions: Biological: Investigational hMPV/RSV vaccine; Biological: Investigational RSV+hMPV vaccine

INTERVENTIONS:
Biological: Investigational hMPV/RSV vaccine — Investigational hMPV/RSV vaccine administered intramuscularly
  Arms: Group 1 Stage 1 Main Cohort; Group 10 Stage 1 Main Cohort; Group 15 Stage 2 Booster Cohort; Group 2 Stage 1 Main Cohort; Group 3 Stage 1 Main Cohort; Group 4 Stage 1 Main Cohort; Group 5 Stage 1 Main Cohort; Group 6 Stage 1 Main Cohort; Group 7 Stage 1 Main Cohort; Group 8 Stage 1 Main Cohort; Group 9 Stage 1 Main Cohort; Group A Stage 1 Sentinel Cohort; Group B Stage 1 Sentinel Cohort; Group X Stage 2 Expansion Cohort
Biological: Investigational hMPV vaccine (monovalent) — Investigational hMPV vaccine (monovalent) administered intramuscularly
  Arms: Group 13 Stage 2 Expansion Cohort
Biological: Investigational RSV vaccine (monovalent) — Investigational RSV vaccine (monovalent) administered intramuscularly
  Arms: Group 12 Stage 2 Expansion Cohort
Biological: Licensed RSV Vaccine — Licensed RSV vaccine administered intramuscularly
  Arms: Group 14 Stage 2 Expansion Cohort
Biological: Placebo — Placebo administered intramuscularly
  Arms: Group 11 Stage 1 Main Cohort; Group C Stage 1 Sentinel Cohort
Biological: Investigational RSV+hMPV vaccine — Investigational RSV+hMPV vaccine administered intramuscularly
  Arms: Group 15 Stage 2 Booster Cohort

SUMMARY:
The aim of this study is to evaluate the safety and immunogenicity of a human metapneumovirus (hMPV) / respiratory syncytial virus (RSV) mRNA vaccine candidate encapsulated in a lipid nanoparticle (LNP) based formulation (hereafter referred to as hMPV/RSV vaccine) for the prevention of lower respiratory tract disease (LRTD) caused by hMPV and/or RSV among adults aged 60 years and older.

The study will also evaluate the safety and immunogenicity of a booster vaccination using a bivalent hMPV/RSV mRNA vaccine candidate (hereafter referred to as RSV+hMPV mRNA vaccine candidate).

Overall, the study is designed to address the following goals:

* Assess the safety profile of the candidate formulations.
* Describe the immunogenicity profile of the candidate formulations.
* Select the vaccine formulations (dose) for future development.
* Assess the safety and immunogenicity of a booster vaccination with the RSV + hMPV mRNA vaccine candidate administered 12 months after primary vaccination with a licensed RSV vaccine.

The study duration is as follows:

-Six months each for the Sentinel and Main Cohorts; up to 12 months for the Expansion Cohort, and 6 additional months for the Booster Cohort

Treatment duration:

* Stage 1 Sentinel Cohort: 1 intra-muscular (IM) injection. Participants will be followed for 6 months post vaccination
* Stage 1 Main Cohort: 1 IM injection. Participants will be followed for 6 months post vaccination
* Stage 2 Expansion Cohort: 1 IM injection. Participants in the licensed RSV vaccine arm will be followed for 12 months post-vaccination; the remainder of the participants will be followed up to 8 months post-vaccination
* Stage 2 Booster Cohort: 1 IM injection 12 months post-primary vaccination. Participants will be followed for 6 months post-booster vaccination

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older on the day of inclusion
* A female participant is eligible to participate if she is not pregnant or breastfeeding and is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year or surgically sterile

Exclusion Criteria:

* Any screening laboratory parameter with laboratory abnormality > Grade 1 deemed clinically significant by the investigator
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months). Of note, persons living with stable human immunodeficiency virus (HIV) are not excluded
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol, polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances; any allergic reaction (eg, anaphylaxis) after administration of an mRNA vaccine
* History of RSV and/or hMPV-associated illness, diagnosed serologically or microbiologically in the last 12 months
* Previous history of myocarditis, pericarditis, and/or myopericarditis
* Screening electrocardiogram that is consistent with possible myocarditis, pericarditis, and/or myopericarditis or, in the opinion of the investigator, demonstrates clinically relevant abnormalities that may affect participant safety or study results
* Laboratory-confirmed thrombocytopenia, contraindicating IM injection, based on investigator's judgment
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection, based on investigator's judgment
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Receipt of any vaccine other than mRNA vaccine in the 28 days preceding any study intervention administration or planned receipt of any vaccine other than mRNA vaccine in the 28 days following any study intervention administration
* Receipt of any mRNA vaccine in the 60 days preceding any study intervention administration or planned receipt of any mRNA vaccine in the 60 days following any study intervention administration
* Previous vaccination against RSV and/or hMPV (with a licensed or investigational vaccine either as a monovalent vaccine or any combination of the antigens)
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1530 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-01-18 (Estimated); Study Completion 2027-01-18 (Estimated)

PRIMARY OUTCOMES:
Presence of unsolicited immediate systemic adverse events (AEs) (Stage 1 and Stage 2 Expansion and Booster Cohorts) | Within 30 minutes after primary and booster vaccinations
  Number of participants reporting immediate unsolicited systemic AEs
Presence of solicited injection site and systemic reactions (Stage 1 and Stage 2 Expansion and Booster Cohorts) | Up to 7 days after primary and booster vaccinations
  Number of participants reporting solicited injection site and systemic reactions
Presence of unsolicited AEs (Stage 1 and Stage 2 Expansion and Booster Cohorts) | Up to 28 days after primary and booster vaccinations
  Number of participants reporting unsolicited AEs
Presence of medically attended AEs (MAAEs) (Stage 1 and Stage 2 Expansion and Booster Cohorts) | Up to 6 months after primary and booster vaccinations
  Number of participants reporting MAAEs
Presence of serious AEs (SAEs) and AEs of special interest (AESIs) (Stage 1 and Stage 2 Expansion and Booster Cohorts) | Up to 6 months after primary and booster vaccinations
  Number of participants reporting SAEs and AESIs
Presence of related SAEs, related AESIs, and fatal SAEs (regardless of causality) (Stage 1 and Stage 2 Expansion and Booster Cohorts) | Throughout the duration of the study (up to approximately 24 months)
  Number of participants reporting related SAEs, related AESIs, and fatal SAEs
Presence of out-of-range biological test results (Stage 1) | Up to 7 days after primary vaccination
  Number of participants with out-of-range biological tests
Presence of out-of-range biological test results (Stage 2 Booster Cohort) | Up to 7 days after booster vaccination
  Number of participants with out-of-range biological tests
hMPV A serum neutralizing antibodies (nAb) titers in Stage 1 Sentinel and Main Cohorts | At pre-vaccination (Day 01) and 28 days post-primary vaccination (Day 29)
  nAb titers expressed as geometric mean titers (GMTs)
hMPV B serum neutralizing antibodies (nAb) titers in Stage 1 Sentinel and Main Cohorts | At pre-vaccination (Day 01) and 28 days post-primary vaccination (Day 29)
  nAb titers expressed as geometric mean titers (GMTs)
RSV A serum nAb titers in Stage 1 Sentinel and Main Cohorts | At pre vaccination (D01) and 28 days post-primary vaccination (D29)
  nAb titers expressed as geometric mean titers (GMTs)
RSV B serum nAb titers in Stage 1 Sentinel and Main Cohorts | At pre vaccination (D01) and 28 days post-primary vaccination (D29)
  nAb titers expressed as geometric mean titers (GMTs)
hMPV A serum neutralizing antibodies (nAb) titers in Stage 2 Expansion Chort | At (Day 01) pre-vaccination and 28 days after the injection of the hMPV/RSV vaccine candidate (Day 29)
  nAb titers expressed as geometric mean titers (GMTs)
hMPV B serum neutralizing antibodies (nAb) titers in Stage 2 Expansion Chort | At (Day 01) pre-vaccination and 28 days after the injection of the hMPV/RSV vaccine candidate (Day 29)
  nAb titers expressed as geometric mean titers (GMTs)
RSV A serum neutralizing antibodies (nAb) titers in Stage 2 Expansion Chort | At (Day 01) pre-vaccination and 28 days after the injection of the hMPV/RSV vaccine candidate (Day 29)
  nAb titers expressed as geometric mean titers (GMTs)
RSV B serum neutralizing antibodies (nAb) titers in Stage 2 Expansion Chort | At (Day 01) pre-vaccination and 28 days after the injection of the hMPV/RSV vaccine candidate (Day 29)
  nAb titers expressed as geometric mean titers (GMTs)
hMPV A serum neutralizing antibodies (nAb) titers in Stage 2 Expansion Chort | At (Day 01) pre-vaccination and 28 days after the injection of the hMPV standalone vaccine (Day 29)
  nAb titers expressed as geometric mean titers (GMTs)
hMPV B serum neutralizing antibodies (nAb) titers in Stage 2 Expansion Chort | At (Day 01) pre-vaccination and 28 days after the injection of the hMPV standalone vaccine (Day 29)
  nAb titers expressed as geometric mean titers (GMTs)
RSV A serum neutralizing antibodies (nAb) titers in Stage 2 Expansion Chort | At (Day 01) pre-vaccination and 28 days after the injection of the RSV standalone vaccine (Day 29)
  nAb titers expressed as geometric mean titers (GMTs)
RSV B serum neutralizing antibodies (nAb) titers in Stage 2 Expansion Chort | At (Day 01) pre-vaccination and 28 days after the injection of the RSV standalone vaccine (Day 29)
  nAb titers expressed as geometric mean titers (GMTs)

SECONDARY OUTCOMES:
hMPV serum anti-F immunoglobulin G (IgG) antibody (Ab) titers (Stage 1) | At pre-vaccination (Day 01) and 28 days (D29) post-primary vaccination
  Ab titers expressed as geometric mean titers (GMTs)
RSV serum anti-F IgG Ab titers (Stage 1) | At pre-vaccination (Day 01) and 28 days (D29) post-primary vaccination
  Ab titers expressed as geometric mean titers (GMTs)
hMPV A serum nAb titers (Stage 2 Expansion Cohort) | At pre-vaccination (Day 01), 28 days (D29), and 3 and 6 months post-primary vaccination
  Ab titers expressed as geometric mean titers (GMTs)
hMPV B serum nAb titers (Stage 2 Expansion Cohort) | At pre-vaccination (Day 01), 28 days (D29), and 3 and 6 months post-primary vaccination
  Ab titers expressed as geometric mean titers (GMTs)
hMPV A serum anti-F IgG Ab titers (Stage 2 Expansion Cohort) | At pre-vaccination (Day 01), 28 days (D29), and 3 and 6 months post-primary vaccination
  Ab titers expressed as geometric mean titers (GMTs)
RSV A serum nAb titers (Stage 2 Expansion Cohort) | At pre-vaccination (Day 01), 28 days (D29), and 3 and 6 months post-primary vaccination
  Ab titers expressed as geometric mean titers (GMTs)
RSV B serum nAb titers (Stage 2 Expansion Cohort) | At pre-vaccination (Day 01), 28 days (D29), and 3 and 6 months post-primary vaccination
  Ab titers expressed as geometric mean titers (GMTs)
RSV serum anti-F IgG Ab titers (Stage 2 Expansion Cohort) | At pre-vaccination (Day 01), 28 days (D29), and 3 and 6 months post-primary vaccination
  Ab titers expressed as geometric mean titers (GMTs)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Velocity Clinical Research, Phoenix- Site Number : 8400025, Phoenix, Arizona
  - CenExel CNS-Garden Grove- Site Number : 8400017, Garden Grove, California
  - National Research Institute - Gardena- Site Number : 8400005, Gardena, California
  - National Research Institute - Huntington Park- Site Number : 8400014, Huntington Park, California
  - Velocity Clinical Research - San Diego- Site Number : 8400008, La Mesa, California
  - Velocity Clinical Research Los Angeles- Site Number : 8400013, Los Angeles, California
  - National Research Institute - Panorama City- Site Number : 8400012, Los Angeles, California
  - Providence Clinical Research - North Hollywood- Site Number : 8400018, North Hollywood, California
  - Peninsula Research Associates- Site Number : 8400002, Rolling Hills Estates, California
  - Velocity Clinical Research - Denver- Site Number : 8400016, Englewood, Colorado
  - Velocity Clinical Research - Washington DC- Site Number : 8400007, Washington D.C., District of Columbia
  - Velocity Clinical Research - Hallandale Beach- Site Number : 8400022, Hallandale, Florida
  - Suncoast Research Associates - Miami - Sunset Drive- Site Number : 8400001, Miami, Florida
  - Velocity Clinical Research - Meridian- Site Number : 8400003, Meridian, Idaho
  - Velocity Clinical Research - Kansas City- Site Number : 8400015, Overland Park, Kansas
  - Velocity Clinical Research - Rockville- Site Number : 8400011, Rockville, Maryland
  - Velocity Clinical Research - Lincoln - Valley Road- Site Number : 8400023, Lincoln, Nebraska
  - Velocity Clinical Research - Omaha- Site Number : 8400006, Omaha, Nebraska
  - Velocity Clinical Research - Springdale- Site Number : 8400004, Cincinnati, Ohio
  - Velocity Clinical Research - Medford- Site Number : 8400024, Medford, Oregon
  - Velocity Clinical Research - Austin- Site Number : 8400020, Cedar Park, Texas
  - Velocity Clinical Research - Salt Lake City- Site Number : 8400010, West Jordan, Utah
  - Velocity Clinical Research - Hampton- Site Number : 8400026, Hampton, Virginia
  - Velocity Clinical Research - Seattle- Site Number : 8400019, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VBD00009 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26215&tenant=MT_SNY_9011